CLINICAL TRIAL: NCT05179876
Title: A Prospective, Open-label, Platform Study for Long-term Follow-up of Participants Using Study Intervention in Pulmonary Hypertension Parent Studies
Brief Title: A Study Providing Treatment Access in Participants With Pulmonary Hypertension Completing a Parent Study and Having no Other Option
Acronym: PLATYPUS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109121; NOPRODPAPUH3001 (Other: Janssen Research & Development, LLC); 2021-002297-11 (EudraCT Number); 2023-506791-27-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-12-17; First posted 2022-01-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hypertension, Pulmonary
Keywords: Chronic thromboembolic pulmonary hypertension (CTEPH); pulmonary arterial hypertension (PAH)
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — macitentan; selexipag

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, extension study, with a platform-study design for long-term safety follow-up of participants using study intervention as in their respective pulmonary hypertension (PH) parent study (that is, pulmonary arterial hypertension [PAH] or chronic thromboembolic pulmonary hypertension [CTEPH]). Participants who have completed a parent study, that benefit from their study intervention maintenance and have no adequate alternative local treatment option (access to the study intervention or an equivalent approved therapy) will be enrolled in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Macitentan (Experimental): Participants who have completed a parent study, benefit from their study intervention maintenance and have no adequate alternative local treatment option will be enrolled in this study and will continue to receive study drug macitentan orally during the course of the study. For adult participants study visits will be scheduled every 6 months and for pediatric participants study visits will be scheduled every 3 months. The study includes on-site visits to collect efficacy and safety information until participant discontinuation/withdrawal, or the respective study intervention is made commercially available in the country/territory or an equivalent approved therapy becomes available, or the sponsor decides to terminate the study prematurely.
  Interventions: Drug: Macitentan
- Selexipag (Experimental): Participants who have completed a parent study, benefit from their study intervention maintenance and have no adequate alternative local treatment option will be enrolled in this study and will continue to receive study drug selexipag orally during the course of the study. Study visits are scheduled every 6 months to collect efficacy and safety information until participant discontinuation/withdrawal, or the respective study intervention is made commercially available in the country/territory or an equivalent approved therapy becomes available, or the sponsor decides to terminate the study prematurely.
  Interventions: Drug: Selexipag
- Macitentan/Tadalafil FDC (Experimental): Participants who have completed a parent study, benefit from their study intervention maintenance and have no adequate alternative local treatment option will be enrolled in this study and will continue to receive drug Macitentan and Tadalafil fixed dose combination (FDC) orally during the course of the study. Study visits are scheduled every 6 months to collect efficacy and safety information until participant discontinuation/withdrawal, or the respective study intervention is made commercially available in the country/territory or an equivalent approved therapy becomes available, or the sponsor decides to terminate the study prematurely.
  Interventions: Drug: Macitentan/Tadalafil FDC

INTERVENTIONS:
Drug: Macitentan — Adult participants will receive oral dose of macitentan 10 milligrams (mg) tablet once daily. Children greater than or equal to (>=) 2 year to less than (<) 18 years will be given an oral macitentan dose tailored to their body weight, ensuring an equivalent level of systemic exposure as in adults.
  Other Names: JNJ-67896062
  Arms: Macitentan
Drug: Selexipag — Adult Participant will receive oral dose of selexipag tablet twice daily at the dose strength corresponding to their maintenance dose at the end of their parent study. Available strengths: 200, 400, 600, 800, 1000, 1200, 1400 and 1600 micrograms (µg). Children with body weight category of >=50 kg will use the tablets at the required dose strength as described for adults. Children with a body weight < 50 kg will receive tablets for pediatric use (dose strengths: 100 and 150 mcg), twice daily to enable continuation of individually maximum tolerated dose of selexipag according to their body weight category.
  Other Names: JNJ-67896049
  Arms: Selexipag
Drug: Macitentan/Tadalafil FDC — Participants will receive oral FDC of macitentan 10 mg and tadalafil 40 mg once daily during the course of the study as already received in the parent studies.
  Other Names: JNJ-68150420
  Arms: Macitentan/Tadalafil FDC

SUMMARY:
The purpose of the study is to enable participants with pulmonary hypertension (PH) currently treated with study intervention(s) in a clinical study (parent studies [NCT03422328, NCT03904693,NCT04565990, NCT02932410, NCT03492177, and NCT04175600]), to continue to benefit from the intervention after closure of the parent study in case they have no alternative means of access to the study intervention. This study will allow assessment of the long-term safety of each study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participant must sign an informed consent form (ICF) (or their legally designated representative must sign) indicating that participant understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Participant treated with oral macitentan or selexipag or fixed dose combination (FDC) of macitentan 10 milligrams (mg) and tadalafil 40 mg at the end of a sponsor parent study and: a) the indication of the parent study is included in the intervention-specific appendices (ISA) (pulmonary arterial hypertension [PAH]; b) participant has completed the parent study; c) no alternative means of access to study intervention (or equivalent approved therapy) have been identified; d) participant may continue to benefit from treatment with the study intervention; e) Participant is at least 18 years old for macitentan/tadalafil FDC, and at least 2 years old for macitentan or selexipag
* A female participant of childbearing potential must: a) have a negative urine or serum pregnancy test prior to first intake of study intervention; b) agree to perform monthly urine pregnancy test up to the end of the safety follow-up period; c) If heterosexually active, agree to follow contraceptive methods until 30 days after the last intake of the study intervention. For pediatric female participants: It is the responsibility of the investigator to ensure appropriate counselling, including consultation with a specialist (if needed), to the participant and/or parent(s)/ legally designated representative (LDR)(s) on the acceptable method of contraception

Exclusion Criteria:

General:

* Participants prematurely discontinued from the study intervention in their parent study
* Female participant being pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study
* Planned or current treatment with another investigational treatment

Macitentan-specific:

* Known allergies, hypersensitivity, or intolerance to macitentan or its excipients
* Hemoglobin less than (<) 80 grams per liter (g/L)
* Serum aspartate (AST) and/or alanine aminotransferases (ALT) greater than (>) 3* upper limit of normal (ULN)
* Known and documented severe hepatic impairment that is, Child-Pugh Class C. For participants with hepatic impairment, Child-Pugh Class (Child-Pugh score) should be fully assessed and documented in the source documents at screening

Selexipag-specific:

* Known allergies, hypersensitivity, or intolerance to selexipag or its excipients
* Suspected or known pulmonary veno-occlusive disease (PVOD)
* Uncontrolled thyroid disease
* Severe coronary heart disease or unstable angina, myocardial infarction within the last 6 months, decompensated cardiac failure (if not under close medical supervision), severe arrhythmia, cerebrovascular events (for example, transient ischemic attack, stroke) within the last 3 months, or congenital or acquired valvular defects with clinically relevant myocardial function disorders not related to pulmonary hypertension (PH)
* Known and documented severe hepatic impairment that is, Child-Pugh Class C. For participants with hepatic impairment, Child-Pugh Class (Child-Pugh score) should be fully assessed and documented in the source documents at screening
* Children only: (a) Current suspicion of intussusception or ileus or gastrointestinal obstruction, per the investigator's judgment; (b) hemoglobin or hematocrit <75 percent (%) of the lower limit of normal range

Macitentan/tadalafil FDC-specific:

* Known allergies, hypersensitivity, or intolerance to macitentan or tadalafil or their excipients
* Hemoglobin <80 g/L
* Serum aspartate (AST) and/or alanine aminotransferases (ALT) >3* ULN range
* Known and documented severe hepatic impairment that is, Child-Pugh Class C. For participants with hepatic impairment, Child-Pugh Class should be fully assessed and documented in the source documents at screening
* Severe renal impairment (estimated glomerular filtration rate [eGF]/creatinine clearance <30 milliliter per minute [mL/min])

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-09-28 (Estimated)

PRIMARY OUTCOMES:
Frequency of Treatment Emergent Adverse Events (TEAEs) | Baseline until End of Study (EOS) (up to 84 months)
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs are defined as a treatment-emergent AE is any AE temporally associated with the use of study treatment (from start of treatment in the PLATYPUS protocol until 30 days after study treatment discontinuation) whether or not considered by the investigator as related to study treatment.
Frequency of TEAEs Leading to Discontinuation | Baseline until EOS (up to 84 months)
  Frequency of TEAEs leading to discontinuation of study intervention will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs are defined as a treatment-emergent AE is any AE temporally associated with the use of study treatment (from start of treatment in the PLATYPUS protocol until 30 days after study treatment discontinuation) whether or not considered by the investigator as related to study treatment.
Frequency of Serious Adverse Events (SAEs) | Baseline until EOS (up to 84 months)
  SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important.
Frequency of Deaths | Baseline until EOS (up to 84 months)
  Frequency of deaths will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Pharmaceuticals Ltd Clinical Trial, Study Director — Actelion
Locations (43):
- Belarus (2):
  - The Republican Scientific-Practical Center ''Cardiology'', Minsk
  - Minsk Regional Clinical Hospital Of The Red Banner Of Labor, Minsk
- UZ Leuven, Leuven, Belgium
- University Multiprofile Hospital for Active Treatment- UMHAT Sveta Anna AD, Sofia, Bulgaria
- China (6):
  - Beijing Anzhen Hospital, Beijing
  - The Second Xiangya Hospital of Central South Hospital, Changsha
  - Jiangsu Province Hospital, Nanjing
  - Qingdao Women and Children's Hospital, Qingdao
  - Childrens Hospital of Shanghai, Shanghai
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- Gottsegen György Országos Kardiológiai Intézet, Budapest, Hungary
- Poland (8):
  - Klinika Kardiologii Z Oddzialem Intensywnego Nadzoru Kardiologicznego UM W Bialymstoku, Bialystok
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Klinika Kardiologii, Bydgoszcz
  - SPSK nr 7 SUM w Katowicach Gornoslaskie Centrum Medyczne im Prof Leszka Gieca, Katowice
  - Oddzial Kardiologii Wojewodzki Szpital Specjalistyczny im W Bieganskiego, Lodz
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego SPZOZ, Lublin
  - SPSK2 PUM Klinika Kardiologii, Szczecin
  - Wojewodzki Szpital Specjalist Osrodek Badawczo Rozwojowy, Wroclaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
- Russia (5):
  - Scientific and Research Institution of Cardiovascular Diseases Complex Problems, Kemerovo
  - E.Meshalkin National Medical Research Center of the Ministry of Health of the Russian Federation, Novosibirsk
  - Federal State Budgetary Institution, Saint Petersburg
  - Institute of Cardiology of Tomsk National Research Medical Center of Rus Academy of Sciences, Tomsk
  - Regional Clinical Hospital No1, Tyumen
- South Africa (2):
  - Abdullah, IA, Durban
  - Dr Kalla, Lenasia
- South Korea (6):
  - Chungnam National University Hospital, Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Taiwan (5):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- Maharaj Nakorn Chiang Mai hospital Faculty of Medicine, Chiang Mai, Thailand
- Ukraine (2):
  - Municipal Inst. Of Dnipropetrovsk Region. Council, Dnipro
  - State Institute Of Phthisiology And Pulmonology N.A. F.G. Yanovskiy Of Ams Ukraine, Kyiv
- Vietnam (3):
  - Hanoi Heart Hospital, Hanoi
  - Hanoi Medical University Hospital, Hanoi
  - Children's Hospital 1, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency